CLINICAL TRIAL: NCT04682977
Title: Piloting the IPROACTIF Program to Preserve Functioning and Prevent Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mansha Parven Mirza, Assoc Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-1461; 5P30AG022849-17 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Heart Disease (Coronary Artery Disease, Ischemic Heart Disease, Hypertensive Heart Disease); Uncontrolled Diabetes (HBA1c ≥ 10)
Keywords: chronic disease; aging; physical function; executive function; activities of daily living; primary care
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Myocardial Ischemia; Chronic Disease | interventions — Occupational Therapy; Aging; Functional Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the IPROACTIF intervention or usual primary care services. Stratified randomization will be carried out with each diagnostic category (diabetes and heart disease) serving as a stratum.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician conducting data analysis will be blinded to group assignment of study participants. A numerical code will be used to identify the study arm for each participant in the outcome database. Outcome measurement will be carried out by blinded assessors at baseline and immediately post-intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPROACTIF (Experimental): 10 weekly sessions. First two sessions focus on comprehensive assessment of physical and executive functioning, assessment of home safety and accessibility, assessment of ADL/IADL competence and performance in context; information in these areas is used by the interventionist to collaboratively identify three patient-centered goals. Goal planning is followed by 10 treatment sessions. Treatment sessions focus on chronic disease education, problem solving issues related to disease management by modifying daily routines, recommendations for embedding physical activity in everyday tasks, and environmental modifications or activity adaptations to increase ADL/IADL independence.
  Interventions: Other: IPROACTIF (Integrated PRimary Care and Occupational Therapy for Aging and Chronic Disease Treatment to preserve Independence and Functioning)
- Usual care (Other): Participants in the control group will receive usual services which might include primary care and prescription medications for chronic disease management.
  Interventions: Other: Usual primary care services

INTERVENTIONS:
Other: IPROACTIF (Integrated PRimary Care and Occupational Therapy for Aging and Chronic Disease Treatment to preserve Independence and Functioning) — IPROACTIF (Integrated PRimary Care and Occupational Therapy for Aging and Chronic Disease Treatment to preserve Independence and Functioning) is an intervention designed to be delivered in primary care settings by an on-site occupational therapist. Based on the premise of preventing the physical and cognitive decline that is associated with aging and chronic disease, the 12-week intervention includes a comprehensive assessment of ADL functioning and ten intervention sessions addressing disease management, physical activity and executive functioning.
  Arms: IPROACTIF
Other: Usual primary care services — Usual primary care services might include monitoring of vitals and other relevant laboratory testing, prescription of medications for chronic disease management, as well as counseling for lifestyle changes.
  Arms: Usual care

SUMMARY:
Conduct a pilot randomized control to assess the preliminary efficacy of IPROACTIF, an occupational therapist-delivered primary care intervention for aging and chronic disease management.

DETAILED DESCRIPTION:
The IPROACTIF intervention is based on the premise of preventing the physical and cognitive decline that is associated with aging and chronic disease. The 12-week intervention includes a comprehensive assessment of ADL functioning and ten intervention sessions addressing disease management, physical activity and executive functioning. This pilot randomized control trial will compare whether patients who receive IPROACTIF perform better than usual care patients on physical functioning, self-efficacy for chronic disease management, physical activity levels, executive functioning, health-related quality of life, and participation in life roles and activities.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Community-dwelling
* 55 years of age
* Primary diagnosis of heart disease (coronary artery disease, ischemic heart disease, hypertensive heart disease), or uncontrolled diabetes (HBA1c greater than/equal to 10)
* Self-reported risk of functional decline (score of 3 or higher) on the 11-item Brief Risk Identification of Geriatric Health Tool or self-reported need for assistance with disease management

Exclusion Criteria

* Current/past diagnosis of stroke or other neurological disorders
* Receiving pharmacological treatment for cognition
* Participating in other exercise or ADL-focused intervention studies
* Non-English speaking
* Residing in a long-term care institution
* Compromised decision-making capacity (score >8 on SOMCT)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mansha Mirza, PhD, OTR/L, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 participants were enrolled. 5 participants who enrolled dropped out/were lost to follow up before randomization to groups. Specifically, these participants began but did not complete all baseline assessments. 40 of the enrolled participants completed all baseline assessments and were assigned to the study arms as indicated in the participant flow.
Period: Overall Study
Arm/Group | IPROACTIF | Usual Care
Started | 18 | 22
Completed | 15 | 20
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPROACTIF | Usual Care | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.0) | 66.7 (7.2) | 66.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 3 | 10 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 13 | 20 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 14 | 25
  White | 4 | 7 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40
Patient-Specific Functional Scale [Mean (Standard Deviation); unit: units on a scale] — The Patient-Specific Functional Scale (PSFS) is a self-reported assessment of activity limitations. Respondents identify up to five important activities they are having difficulty with because of their health condition. Each activity is rated on a scale from 0 (unable to perform) to 10 (able to perform at same level as before). Total score is the sum of the activity scores/number of activities and can range from 0 to 10. Higher score indicates a better outcome.
  units on a scale | 5.81 (2.08) | 4.92 (1.63) | 5.32 (1.88)
PROMIS Physical Function Short Form 20 [Mean (Standard Deviation); unit: T-score] — The PROMIS Physical Function Short Form 20 (PF-20) is a measure of perceived ability to perform physical activities. Respondents rate 20 daily activities on a scale from 1 (unable to do) to 5 (no difficulty/limitation). Individual item scores are summed to compute the total raw score which is converted to a standardized T-score. T-scores range from 9.2 to 62.7.
  Higher T-scores indicate a better outcome. A score of 50 is the average for the United States general population with a standard deviation of 10.
  T-score | 41.12 (7.64) | 40.12 (8.65) | 40.57 (1.88)
Physical Performance Test [Mean (Standard Deviation); unit: units on a scale] — The Physical Performance Test (PPT) is an assessment of physical function based on directly observed performance of nine tasks that simulate daily living activities. Each task is scored on a scale ranging from 0 (unable to do) to 4 (most capable or fastest) and scores are summed to generate a total score. Scores range from 0 to 36. Higher score indicates a better outcome.
  units on a scale | 24.50 (6.38) | 24.18 (7.30) | 24.33 (6.82)
Exercise Regularly Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 3 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 7.15 [2.7 to 10] | 6.70 [2.3 to 10] | 6.70 [2.3 to 10]
Obtain Help from Community, Family, Friends Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 4 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 7.8 [2.8 to 10] | 7 [2 to 10] | 7.4 [2 to 10]
Manage Disease in General Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 5 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 8.2 [6.8 to 10] | 7.8 [3.6 to 10] | 8 [3.6 to 10]
Social Recreational Activities Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 2 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 7.75 [4.0 to 10] | 7.5 [2.5 to 10] | 7.5 [2.5 to 10]
Doing Chores Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 3 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 8.15 [3 to 10] | 7 [2 to 10] | 7.85 [2 to 10]
Manage Symptoms Scale from the Self-Management Resource Center [Median (Full Range); unit: units on a scale] — This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 5 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
  units on a scale | 7.1 [3.6 to 9] | 6.2 [2.6 to 10] | 6.7 [2.6 to 10]
Late Life Functioning and Disability Index (Disability Component) - Frequency Dimension [Mean (Standard Deviation); unit: units on a scale] — The Late Life Function and Disability Inventory (LLFDI, Disability Component) measures participation in major life activities and roles. For the frequency dimension, respondents rate how often they perform each activity on a scale from 1 (never) to 5 (very often). Individual item scores are summed to compute the total raw score for the frequency dimension. Raw scores are then converted to a standardized scale score. Scale scores range from o to 100. Higher score indicates a better outcome.
  units on a scale | 48.94 (5.64) | 49.48 (8.55) | 49.24 (7.30)
Late Life Functioning and Disability Index (Disability Component)- Limitations Dimension [Mean (Standard Deviation); unit: units on a scale] — The Late Life Function and Disability Inventory (LLFDI, Disability Component) measures participation in major life activities and roles. For the limitations dimension, respondents rate how limited they feel in completing each activity on a scale from 1 (completely) to 5 (not at all). Individual item scores are summed to compute the total raw score for the limitations dimension. Raw scores are then converted to a standardized scale score. Scale scores range from o to 100. Higher score indicates a better outcome.
  units on a scale | 66.26 (10.04) | 66.62 (16.98) | 66.46 (14.12)
PROMIS Global Health Measure (physical subscale) [Mean (Standard Deviation); unit: T-score] — The PROMIS Global Health Short Form is a 10-item self-report assessment of health-related quality of life (HRQOL). Item scores are summed to compute raw scores for physical and mental health. Raw scores are converted to T-scores using a standard conversion table. T-scores for the physical health sub-scale range from 16.2 to 67.7.
  A T-Score of 50 represents the average (mean) for the US general population with a standard deviation of 10 points.
  Higher T-scores indicate a better outcome.
  T-score | 42.36 (8.37) | 42.14 (8.91) | 42.24 (8.56)
PROMIS Global Health Measure (mental subscale) [Mean (Standard Deviation); unit: T-score] — The PROMIS Global Health Short Form is a 10-item self-report assessment of health-related quality of life (HRQOL). Item scores are summed to compute raw scores for physical and mental health. Raw scores are converted to T-scores using a standard conversion table. T-scores for the mental health sub-scale range from 21.2 to 67.6.
  A T-Score of 50 represents the average (mean) for the US general population with a standard deviation of 10 points.
  Higher T-scores indicate a better outcome.
  T-score | 44.88 (7.40) | 45.53 (8.75) | 45.24 (8.08)
Executive Function Performance Test [Median (Full Range); unit: units on a scale] — The Executive Function Performance Test (EFOT) is a performance-based assessment of an individual's executive functioning abilities in the context of a specific task. The original assessment comprises three tasks; only the medication management task was used in this study. Scores range from 0-25 for this task. Higher scores indicate poorer performance.
  units on a scale | 4.5 [0 to 13] | 4 [0 to 12] | 4 [0 to 13]
Performance Assessment of Self-care Skills [Median (Full Range); unit: units on a scale] — The Performance Assessment of Self-care Skills (PASS) is a performance-based assessment on and individual's ability to perform ADL/IADL tasks safely and independently. The individual is expected to perform an ADL/IADL task which is rated on independence, safety, and adequacy. Independence scores range from 0-3; higher scores indicate better performance.
  units on a scale | 2.92 [1.00 to 3.00] | 3 [0.67 to 3.00] | 3 [0.67 to 3.00]
Average time spent in moderate to vigorous physical activity (accelerometry) [Median (Full Range); unit: minutes] — Average time spent in moderate to vigorous physical activity as measured by an accelerometer worn for at least 6 hours for at least 4 days during a 7-day period. This is not a scale measure. Higher number indicates greater level of physical activity. Population: Number analyzed is lower than the overall number for each group due to missing data. Not all participants returned the accelerometer with valid and usable data.
  minutes
    number analyzed (Participants) | 17 | 19 | 36
    (all) | 4.21 [1.57 to 87.86] | 5.04 [0.50 to 56] | 4.35 [0.50 to 87.86]
Dimensional Change Card Sort [Median (Full Range); unit: units on a scale] — The NIH Toolbox Dimensional Change Card Sort (DCCS) Test is a computer-administered measure of cognitive flexibility and attention. Test takers match bivalent test pictures to the target pictures along dimensions of shape and color. Scoring is based on combining accuracy and reaction time & converted to a scale score with mean of 100 and SD of 15. Scale scores may be adjusted for age. Adjusted scores are relative to a normative sample with no universally applicable fixed minimum or maximum. Higher scores indicate better performance.
  Scores listed represent unadjusted scale scores.
  units on a scale | 95 [51 to 103] | 95 [51 to 109] | 95 [51 to 109]

OUTCOME MEASURES:

1. Primary Outcome: Physical Functioning Measured Using the Patient-Specific Functional Scale
Description: Validated self-reported assessment; respondent identifies up to 5 important activities they are experiencing difficulty with. Total score = sum of the activity scores/number of activities. scoring Scores can range from 0 to 10; higher scores indicate better physical functioning
  Minimal clinically important difference in previous studies = 1.2-2.2 points
Time Frame: 12 weeks
Population: Intent to Treat population (all participants assigned to IPROACTIF or Control). Expectation Maximization imputation method.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 7.45 (2.64) | 5.43 (2.31)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.04, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 1.58, Standard Error of Mean 0.76 — Treatment Difference = IPROACTIF-Control

2. Primary Outcome: Physical Functioning Measured Using the PROMIS Physical Function Short Form 20
Description: The PROMIS Physical Function Short Form 20 (PF-20) is a measure of perceived ability to perform physical activities. Respondents rate 20 daily activities on a scale from 1 (unable to do) to 5 (no difficulty/limitation). Individual item scores are summed to compute the total raw score which is converted to a standardized T-score. T-scores range from 9.2 to 62.7.
  Higher T-scores indicate a better outcome. A score of 50 is the average for the United States general population with a standard deviation of 10.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
units on a scale | 43.91 (12.06) | 40.79 (9.69)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.26, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 1.98, Standard Error of Mean 1.75 — Treatment Difference = IPROACTIF-Control

3. Primary Outcome: Physical Functioning Measured Using the Physical Performance Test (9-item)
Description: 9-item performance-based assessment; scores can range from 0 to 36; higher scores indicate better physical functioning Minimal clinically important difference in previous studies = 2.4 points
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 24.7 (8.73) | 25.4 (6.42)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.51, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = -1.06, Standard Error of Mean 1.60 — Treatment Difference = IPROACTIF-Control

4. Secondary Outcome: Participation in Life Activities and Roles Using the Late Life Functioning and Disability Index (Disability Component) - Frequency Dimension
Description: 16-item self-reported measure; scaled scores for the frequency dimension range from 0-100; higher scores indicate greater frequency i.e. better performance.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 52.01 (7.02) | 50.30 (9.39)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.23, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 2.17, Standard Error of Mean 1.78 — Treatment Difference = IPROACTIF - Control

5. Secondary Outcome: Participation in Life Activities and Roles Using the Late Life Functioning and Disability Index (Disability Component) - Limitations Dimension
Description: 16-item self-reported measure; scaled scores for the frequency dimension range from 0-100; higher scores indicate lesser difficulty i.e. better performance.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 74.70 (26.17) | 70.41 (21.03)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.44, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 4.65, Standard Error of Mean 5.97 — Treatment Difference = IPROACTIF - Control

6. Secondary Outcome: Health Related Quality of Life Using the PROMIS Global Health Measure (Physical Subscale)
Description: The PROMIS Global Health Short Form is a 10-item self-report assessment of health-related quality of life (HRQOL). Item scores are summed to compute raw scores for physical and mental health. Raw scores are converted to T-scores using a standard conversion table. T-scores for the physical health sub-scale range from 16.2 to 67.7.
  A T-Score of 50 represents the average (mean) for the US general population with a standard deviation of 10 points.
  Higher T-scores indicate a better outcome.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 48.36 (15.90) | 43.21 (8.89)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.22, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 4.37, Standard Error of Mean 3.47 — Treatment Difference = IPROACTIF - Control

7. Secondary Outcome: Health Related Quality of Life Using the PROMIS Global Health Measure (Mental Subscale)
Description: The PROMIS Global Health Short Form is a 10-item self-report assessment of health-related quality of life (HRQOL). Item scores are summed to compute raw scores for physical and mental health. Raw scores are converted to T-scores using a standard conversion table. T-scores for the mental health sub-scale range from 21.2 to 67.6.
  A T-Score of 50 represents the average (mean) for the US general population with a standard deviation of 10 points.
  Higher T-scores indicate a better outcome.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 45.71 (8.23) | 46.38 (7.93)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.91, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 0.91, Standard Error of Mean 1.80 — Treatment Difference = IPROACTIF - Control

8. Secondary Outcome: Self-efficacy Measured Using the Doing Chores Scale From the Self-Management Resource Center
Description: This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 3 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 8.14 (2.36) | 6.98 (3.04)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.78, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = 0.18, Standard Error of Mean 0.65 — Treatment Difference = IPROACTIF - Control

9. Secondary Outcome: Self-efficacy Measured Using the Manage Symptoms Scale From the Self-Management Resource Center
Description: This is a scale within the Chronic Disease Self-Efficacy Scales (CDSES) measure which assesses perceived confidence for performing specific behaviors for managing chronic health conditions and their sequelae. This scale includes 5 items. Items are rated on a scale of 1 (not at all confident) to 10 (totally confident). The total scale score is the mean of the items and can range from 1 to 10. Higher score indicates a better outcome.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 7.30 (2.05) | 7.18 (2.21)
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.83, ANCOVA — Sidak correction for multiple comparisons; ANCOVA with baseline score as covariate Effect size calculated using Cohen's d; Mean difference (adjusted) = -0.12, Standard Error of Mean 0.53 — Treatment Difference = IPROACTIF - Control

10. Secondary Outcome: Self-efficacy for Chronic Disease Management Using the Obtain Help From Community, Family, Friends Scale From the Self-Management Resource Center
Description: Change from pre-test (baseline) to post-test (12 weeks) in self-efficacy for getting support from others as measured on a 4-item validated self-reported assessment; Scores range from 1 to 10; higher scores indicate better self-efficacy
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 0.10 [-3.30 to 5.30] | 0.35 [-2.80 to 4.20]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.67, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; A non-parametric test was used due to non-normal distribution of data. Effect size calculated using rank biserial correlation r

11. Secondary Outcome: Self-efficacy for Chronic Disease Management Using the Manage Disease in General Scale From the Self-Management Resource Center
Description: Change from pre-test (baseline) to post-test (12 weeks) in self-efficacy for general disease management as measured on a 5-item validated self-reported assessment; Scores range from 1 to 10; higher scores indicate better self-efficacy
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 0.20 [-3.88 to 3.20] | 0.00 [-4.20 to 3.00]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Self-efficacy for Chronic Disease Management Using the Social Recreational Activities Scale From the Self-Management Resource Center
Description: Change from pre-test (baseline) to post-test (12 weeks) in self-efficacy for engaging in social and recreational activities as measured on a 2-item validated self-reported assessment; Scores range from 1 to 10; higher scores indicate better self-efficacy
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 0.02 [-2.50 to 5.00] | 0.50 [-5.00 to 3.04]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

13. Secondary Outcome: Self-efficacy for Chronic Disease Management Using the Exercise Regularly Scale From the Self-Management Resource Center
Description: Change from pre-test (baseline) to post-test (12 weeks) in self-efficacy for getting regular exercise as measured on a 3-item validated self-reported assessment; scores range from 1 to 10; higher scores indicate better self-efficacy
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 1.02 [-2.40 to 6.30] | 0.24 [-3.70 to 5.00]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

14. Secondary Outcome: Performance of Daily Living Tasks Using the Performance Assessment of Self-care Skills
Description: Change from pre-test (baseline) to post-test (12 weeks) as measured on the Performance Assessment of Self-care Skills (PASS). The PASS is a performance-based assessment; individual is expected to perform an ADL/IADL task which is rated on independence, safety, and adequacy. Independence scores range from 0-3; higher scores indicate better performance
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 0.09 [-1.6 to 1.5] | 0.00 [-0.69 to 2.17]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

15. Secondary Outcome: Executive Functioning Using the Executive Function Performance Test
Description: Change from pre-test (baseline) to post-test (12 weeks) as measured on the Executive Function Performance Test (EFPT). The EFPT is a performance-based assessment; original assessment comprises three tasks; only the medication management task was used; scores range from 0-25 for this task; higher scores indicate poorer performance.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 1.70 [-9.00 to 7.00] | 1.00 [-6.00 to 7.00]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

16. Secondary Outcome: Executive Functioning Using the Dimensional Change Card Sort Test
Description: The NIH Toolbox Dimensional Change Card Sort (DCCS) Test is a computer-administered measure of cognitive flexibility and attention. Test takers match bivalent test pictures to the target pictures along dimensions of shape and color. Scoring is based on combining accuracy and reaction time & converted to a scale score with mean of 100 and SD of 15. Scale scores may be adjusted for age. Adjusted scores are relative to a normative sample with no universally applicable fixed minimum or maximum. Higher scores indicate better performance.
  Scores listed represent unadjusted scale scores.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 18 | 22
score on a scale | 4.00 [-36.00 to 18.87] | 3.94 [-7.00 to 32.00]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.81, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

17. Secondary Outcome: Physical Activity Level
Description: Change from pre-test (baseline) to post-test (12 weeks) in the average time spent in moderate to vigorous physical activity as measured by an accelerometer worn for at least 6 hours for at least 4 days during a 7-day period.
Time Frame: 12 weeks
Population: Intent to Treat population (all participants assigned to IPROACTIF or Control).
Measure: Median (Full Range); unit: minutes
Arm/Group | IPROACTIF | Usual Care
Number analyzed (Participants) | 13 | 15
minutes | -0.85 [-60.07 to 10.71] | 0.07 [-12.36 to 15.64]
Statistical Analysis 1: Comparison: IPROACTIF vs Usual Care; Test type: Superiority; p = 0.89, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | IPROACTIF | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 1/18 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPROACTIF (N=18) | Usual Care (N=22)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — The participant had a fall when walking to the study lab. She did not sustain serious injury. The PI followed up with her daily for a week; no further concerns were reported. The incident was reported to the IRB and deemed unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT04682977/Prot_SAP_000.pdf